CLINICAL TRIAL: NCT03215420
Title: Diagnostic Agreement of Electrophysiological Audiovestibular Examinations With Magnetic Resonance Imaging (MRI) of the Inner Ear in Revealing Endolymphatic Hydrops (EH) in Patients With Certain or Probable Meniere's Disease (MD)
Brief Title: Comparison of 3 Methods to Diagnose Endolymphatic Hydrops in Meniere's Disease
Acronym: MRI Meniere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DIORFLAR- BOZORG 2016
Record Dates: First submitted 2017-06-26; First posted 2017-07-12 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Endolymphatic Hydrops
MeSH Terms: conditions — Endolymphatic Hydrops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Certain or probable Meniere's disease (Experimental)
  Interventions: Diagnostic Test: MRI 3T

INTERVENTIONS:
Diagnostic Test: MRI 3T

SUMMARY:
The aim of this study is to compare 3 methods for the diagnosis of endolymphatic hydrops (EH) in patients with Meniere's disease: MRI 3 Tesla (to visualise EH directly), and functional explorations, namely electrocochleography and dephasing of acoustic distortion products (which are modified by the EH).

The research hypothesis is that the examinations will show agreement in the diagnosis of EH, and that the results obtained (quantitative values) will vary in the same direction over time and during flares of MD.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written consent
* persons aged 18 to 75 years
* persons with certain, probable or possible Meniere's disease according to the international classification AAO-HNS

Exclusion Criteria:

* persons without health insurance cover
* adults under guardianship
* persons with a history of hypersensitivity to the active substance or to one of the excipients of the contrast agent used for the MRI or to any gadolinium chelate
* pregnant or breast-feeding women
* severe acute or chronic kidney failure
* other identified causes of cochleo-vestibular syndromes
* Impossibility to follow-up or carry out any of the examinations necessary for the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Number of patients for whom an endolymphatic hydrops was diagnosed by electrocochleography | day one
Number of patients for whom an endolymphatic hydrops was diagnosed by (Dephasing) of acoustic distortion products | day one
Number of patients for whom an endolymphatic hydrops was diagnosed by 3T MRI 3T | day one

CONTACTS AND LOCATIONS:
Locations (1):
- CHu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No